CLINICAL TRIAL: NCT04018820
Title: Effects of a 12-week Strength Training Program in Men With Myotonic Dystrophy Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Élise Duchesne (Other)
Collaborators: Fondation du Grand défi Pierre Lavoie (Unknown)
Responsible Party: Sponsor-Investigator, Élise Duchesne, Sponsor-Investigator, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-005
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Intervention Model Description: Participants had to complete a 12-week strength training program and return to their normal activities for the following 6 months after the end of the training program
Masking Description: Most outcomes where not masked, however the outcome assessor was masked for all muscle biopsy analysis: while analysing the muscle biopsy outcomes, the outcome assessor did not know if it was from baseline or from after the training program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training program (Experimental)
  Interventions: Other: Training program

INTERVENTIONS:
Other: Training program — 12-week strength training program of the lower limbs consisting of 5 different exercises: Leg extension, leg press, hip abduction, squat and plantar flexion. All exercises were performed between 6 and 8 maximal repetitions.

SUMMARY:
Eleven men with myotonic dystrophy type 1 (DM1) underwent a 12-week lower-limb strength training program. The training program consisted of 3 series of 6 to 8 maximal repetitions of 5 different exercises: Leg extension, leg press, hip abduction, squat and plantar flexion. Training sessions were closely supervised and took place twice a week. It is hypothesised that the training program will induce muscular hypertrophy despite the genetic defect. The training program should also have positive effects on function. The participants were evaluated at baseline, week 6, week 12, month 6 and month 9 to see the effects of the training program and if these effects are maintained over time.

ELIGIBILITY:
Inclusion Criteria:

* DM1 diagnosis must be confirmed by genetic analysis;
* Male gender, aged between 30 and 65 years old;
* Be able to walk without assistance;
* Consent of the neurologist must be given to participate in this study;
* Must reside in the Saguenay-Lac-St-Jean region;
* Subjects must be able to give their consent freely and voluntarily.

Exclusion Criteria:

* Patients with any other form of muscular dystrophy are excluded;
* Any contraindication for strenuous exercise or muscle biopsy.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Changes in maximal isometric muscle strength of the knee extensors | At baseline, week 6, week 12, month 6 and month 9
  Changes in maximal isometric muscle strength of the knee extensors measured by quantified muscle testing using a handheld dynamometer

SECONDARY OUTCOMES:
Changes in maximal isometric muscle strength of the knee flexors | At baseline and week 12
  Changes in maximal isometric muscle strength of the knee flexors measured by quantified muscle testing using a handheld dynamometer
Changes in maximal isometric muscle strength of the hip flexors | At baseline and week 12
  Changes in maximal isometric muscle strength of the hip flexors measured by quantified muscle testing using a handheld dynamometer
Changes in maximal isometric muscle strength of the hip extensors | At baseline and week 12
  Changes in maximal isometric muscle strength of the hip extensors measured by quantified muscle testing using a handheld dynamometer
Changes in maximal isometric muscle strength of the ankle dorsiflexors | At baseline and week 12
  Changes in maximal isometric muscle strength of the ankle dorsiflexors measured by quantified muscle testing using a handheld dynamometer
Changes in 1-repetition maximum strength of the leg extension exercise | At baseline, week 6 and week 12
  Changes in 1-repetition maximum strength of the leg extension exercise
Changes in 1-repetition maximum strength of the leg press exercise | At baseline, week 6 and week 12
  Changes in 1-repetition maximum strength of the leg press exercise
Changes in 1-repetition maximum strength of the hip abduction exercise | At baseline, week 6 and week 12
  Changes in 1-repetition maximum strength of the hip abduction exercise
Changes in 1-repetition maximum strength of the squat exercise | At baseline, week 6 and week 12
  Changes in 1-repetition maximum strength of the squat exercise
Changes in comfortable walking speed in the 10-meter walk test | At baseline, week 6, week 12, month 6 and month 9
  Changes in comfortable walking speed in the 10-meter walk test
Changes in maximal walking speed in the 10-meter walk test | At baseline, week 6, week 12, month 6 and month 9
  Changes in maximal walking speed in the 10-meter walk test
Changes in the number of repetitions in the 30-seconds sit-to-stand test | At baseline, week 6, week 12, month 6 and month 9
  Changes in the number of repetitions in the 30-seconds sit-to-stand test
Changes in the score of the lower extremity functional scale | At baseline, week 12, month 6 and month 9
  Changes in the score of the lower extremity functional scale (LEFS). The LEFS is an 80-point questionnaire with 20 items scored from 0 to 4. A score of 80 means no disfunction while a score of 0 means maximal disfunction.
Changes in the score of the myotonic dystrophy health index | At baseline, week 6, week 12, month 6 and month 9
  Changes in the score of the myotonic dystrophy health index (MDHI). The MDHI is a 114-item questionnaire scored from 0 to 100, where 0 means no disability and 100 means maximal disability.
Changes in the score of the Fatigue and Daytime Sleepiness Scale | At baseline, week 6, week 12, month 6 and month 9
  Changes in the score of the Fatigue and Daytime Sleepiness Scale (FDSS). The FDSS is a 12-item questionnaire where all questions are scored from 0 to 2. A higher score means more daytime sleepiness and fatigue.
Changes in the Marin apathy scale | At baseline, week 12, month 6 and month 9
  Changes in the Marin apathy scale. The Marin apathy scale is scored by the clinician where he interviews the subject and then scores an 18-item list on a scale of 1 to 4. A high score means more apathy.
Changes in the Well-Being Manifestations Measure Scale | At baseline, week 6, week 12 and month 6
  Changes in the Well-Being Manifestations Measure Scale (WBMMS). The WBMMS is a 25-item questionnaire where each question is scored on a scale from 1 to 5. A high score means high well-being.
Changes in the Hospital Anxiety and Depression Scale | At baseline, week 6, week 12 and month 6
  Changes in the Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item questionnaire with a scale from 0 to 3 for each item. A high score means high depression and anxiety.
Changes in muscle biopsy of the vastus lateralis: muscle fiber typing | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: muscle fiber typing
Changes in muscle biopsy of the vastus lateralis: muscle fiber size | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: muscle fiber size (smallest diameter of the fiber)
Changes in muscle biopsy of the vastus lateralis: muscle proteomics | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: muscle proteomics (protein expression)
Changes in muscle biopsy of the vastus lateralis: muscle transcriptomics | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: muscle transcriptomics (RNA expression analysis)
Changes in muscle biopsy of the vastus lateralis: mitochondrial function | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: mitochondrial function. Analysis of mitochondrial markers and enzymes
Changes in muscle biopsy of the vastus lateralis: Nuclear foci | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: Nuclear foci (changes in accumulation of nuclear foci)

CONTACTS AND LOCATIONS:
Overall Officials: Elise Duchesne, Ph.D., Principal Investigator — Université du Québec à Chicoutimi
Locations (1):
- Groupe de recherche interdisciplinaire sur les maladies neuromusculaires, Saguenay, Quebec, Canada